CLINICAL TRIAL: NCT01039818
Title: Comparison of Different Doses of 131I in Severe Graves' Hyperthyroidism: A Clinical Trial With Historical Control
Brief Title: Comparison of Different Doses of 131I in Severe Graves' Hyperthyroidism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Ana Luiza Maia, PhD, Hospital de Clinicas de Porto Alegre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-055
Record Dates: First submitted 2009-12-24; First posted 2009-12-25 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-09

CONDITIONS: Graves Disease
Keywords: Graves Disease; Hyperthyroidism; Radioiodine; Clinical trial
MeSH Terms: conditions — Graves Disease; Hyperthyroidism | interventions — Iodine-131

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiodine-200µCi (Active Comparator): A subgroup of patients with Graves' Disease and goiter ≥48ml treated with 200µCi of ¹³¹I/ml thyroid tissue, corrected by 24h-RAIU, from a randomized controlled trial run at our institution between February 1997 and March 2000, serves as a historical control.
  Interventions: Radiation: Radioiodine
- Radiodine-250µCi (Experimental): Patients with Graves' Disease and goiter ≥48ml, prospectively assigned to receive 250 µCi of ¹³¹I/ml thyroid tissue, corrected by 24h-RAIU.
  Interventions: Radiation: Radioiodine

INTERVENTIONS:
Radiation: Radioiodine — A unique dose of 200µCi of ¹³¹I/ml/24-RAIU
  Arms: Radiodine-200µCi
Radiation: Radioiodine — A unique dose of 250µCi of ¹³¹I/ml/24-RAIU
  Arms: Radiodine-250µCi

SUMMARY:
The purpose of this study is to determine whether higher doses of radioiodine increase treatment efficacy in severe Graves' disease.

DETAILED DESCRIPTION:
Graves' disease (GD) is the most frequent cause of hyperthyroidism, affecting mainly women aged 40-60 years. Radioiodine (¹³¹I), introduced in 1941, has become a cornerstone in the treatment of GD hyperthyroidism. Because of its safety, low costs and rapid effect, it is considered a first line therapy in the United States. However, treatment failure occurs in about 15-25% of patients treated with radioiodine. Patients not cured with the first dose of radioiodine usually present severe hyperthyroidism, characterized by large goiter, high 24-hour radioiodine uptake (24h-RAIU) and very high levels of thyroid hormones. We have previously shown that large goiter (≥48ml) is an independent predictor of treatment failure. In these patients, the therapeutic failure was 40.0% while in patients with smaller goiter was only 6.5% (P=0.005; unpublished). It is generally accepted that higher doses of radioiodine improves cure rates. Indeed, a recent meta-analysis found a correlation between radioiodine dose and therapeutic success in GD patients. To our knowledge, there are no published studies evaluating cure rates with different radioiodine doses in severe GD.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with a recent diagnosis of Graves' disease and goiter ≥ 48 ml, attending the Endocrine Division at Hospital de Clinicas de Porto Alegre are eligible.

Exclusion Criteria:

* Patients with previous treatment with radioiodine or thyroidectomy,
* Signs of moderate or severe ophthalmopathy (proptosis > 22 mm, ophthalmoplegia, chemosis, or lagophthalmos),
* Severe heart disease (symptomatic coronary heart disease, class III heart failure, New York Heart Association criteria),
* Debilitating conditions, and
* Large and compressive goiters (> 150 g).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 1997-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Cure, defined as euthyroidism or permanent hypothyroidism based on FT4 measurements. | 12 months

SECONDARY OUTCOMES:
Euthyroidism | 12 months
Permanent hypothyroidism | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ana L Maia, MD, PhD, Principal Investigator — Thyroid Unit, Endocrine Division, Hospital de Clínicas de Porto Alegre
Locations (1):
- Thyroid Unit, Endocrine Division, Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Andrade VA, Gross JL, Maia AL. Effect of methimazole pretreatment on serum thyroid hormone levels after radioactive treatment in Graves' hyperthyroidism. J Clin Endocrinol Metab. 1999 Nov;84(11):4012-6. doi: 10.1210/jcem.84.11.6149. PMID 10566642
- [Background] Andrade VA, Gross JL, Maia AL. The effect of methimazole pretreatment on the efficacy of radioactive iodine therapy in Graves' hyperthyroidism: one-year follow-up of a prospective, randomized study. J Clin Endocrinol Metab. 2001 Aug;86(8):3488-93. doi: 10.1210/jcem.86.8.7707. PMID 11502768
- [Background] Andrade VA, Gross JL, Maia AL. Serum thyrotropin-receptor autoantibodies levels after I therapy in Graves' patients: effect of pretreatment with methimazole evaluated by a prospective, randomized study. Eur J Endocrinol. 2004 Oct;151(4):467-74. doi: 10.1530/eje.0.1510467. PMID 15476447
- [Background] Andrade VA, Gross JL, Maia AL. [Radioactive iodine therapy in Graves' hyperthyroidism]. Arq Bras Endocrinol Metabol. 2004 Feb;48(1):159-65. doi: 10.1590/s0004-27302004000100017. Epub 2004 Jun 1. Portuguese. PMID 15611828
- [Derived] Dora JM, Escouto Machado W, Andrade VA, Scheffel RS, Maia AL. Increasing the radioiodine dose does not improve cure rates in severe graves' hyperthyroidism: a clinical trial with historical control. J Thyroid Res. 2013;2013:958276. doi: 10.1155/2013/958276. Epub 2013 Jul 31. PMID 23984185